CLINICAL TRIAL: NCT01460888
Title: Radiotherapy & Olaparib in COmbination for Carcinoma of the Oesophagus. A Phase I Trial.
Brief Title: Radiotherapy & Olaparib in COmbination for Carcinoma of the Oesophagus
Acronym: ROCOCO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10_DOG03_194
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2011-12

CONDITIONS: Carcinoma of the Oesophagus
MeSH Terms: conditions — Esophageal Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- OLA-0 (de-escalation dose) (Experimental): 25mg olaparib twice daily + radiotherapy (50Gy in 25 fractions)
  Interventions: Drug: Olaparib; Radiation: Radical external beam radiotherapy, 50Gy in 25 fractions
- OLA-1 (Experimental): 50mg olaparib twice daily + radiotherapy (50Gy in 25 fractions)
  Interventions: Drug: Olaparib; Radiation: Radical external beam radiotherapy, 50Gy in 25 fractions
- OLA-2 (Experimental): 100mg olaparib twice daily + radiotherapy (50Gy in 25 fractions)
  Interventions: Drug: Olaparib; Radiation: Radical external beam radiotherapy, 50Gy in 25 fractions
- OLA-3 (Experimental): 200mg olaparib twice daily + radiotherapy (50Gy in 25 fractions)
  Interventions: Drug: Olaparib; Radiation: Radical external beam radiotherapy, 50Gy in 25 fractions
- RT alone (Active Comparator)
  Interventions: Radiation: Radical external beam radiotherapy, 50Gy in 25 fractions

INTERVENTIONS:
Drug: Olaparib — 25mg tablets, oral. Commenced 3 days prior to radiotherapy and continuing until the last day of radiotherapy (36 days in total).
  Arms: OLA-0 (de-escalation dose); OLA-1; OLA-2; OLA-3
Radiation: Radical external beam radiotherapy, 50Gy in 25 fractions — Radiotherapy to the oesophageal carcinoma. For patients receiving olaparib this is delivered as 50Gy in 25 daily fractions for 5 weeks (Monday-Friday only). For patients in the comparator arm (RT only) other total doses/ fractionation are permitted, according to local policy/ best standard care.

SUMMARY:
The purpose of this study is to determine the Maximum Tolerated Dose (MTD) of olaparib in combination with radical radiotherapy in patients with oesophageal cancer who are unsuitable for platinum containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma or squamous cell carcinoma of the oesophagus including Siewert type 1 or 2 tumours with ≤2cm gastric mucosal extension
2. Unsuitable for radical chemoradiation therapy but suitable for radiotherapy
3. Total length of tumour and involved lymph nodes ≤10cm
4. No oesophageal stent in situ
5. No previous chemotherapy or radiotherapy for oesophagus cancer
6. Disease which can be encompassed within a radical radiotherapy treatment volume
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (see ECOG criteria appendix 1)
8. Provision of fully informed consent, signed, written and dated, prior to any study specific procedures.
9. > 18 years of age.
10. Adequate organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥ 10.0 g/dL
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * White blood cells (WBC) > 3 x 109/L
    * Platelet count ≥ 100 x 109/L
    * No dysplastic features on peripheral blood smear
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal
    * Aspartate aminotransferase (AST(SGOT)/Alanine transaminase (ALT)SGPT) ≤ 2.5 x institutional upper limit of normal
    * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN)
11. Adequate lung function: no history of interstitial lung disease and FEV1 > 1litre and >30% predicted.
12. Evidence of non-childbearing status for women of childbearing potential, or postmenopausal status: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. Postmenopausal is defined as:

    * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    * Luteinizing hormone(LH) and Follicle-stimulating hormone (FSH) levels in the post menopausal range for women under 50,
    * radiation-induced oophorectomy with last menses >1 year ago,
    * chemotherapy-induced menopause with >1 year interval since last menses,
    * surgical sterilisation (bilateral oophorectomy or hysterectomy).
13. Patient willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
14. Fit to receive all study treatments
15. Swallowing sufficiently good to tolerate oral medication
16. Life expectancy ≥ 4 months.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Treatment with any investigational product during the last 14 days (or a longer period depending on the defined characteristics of the agents used)
4. Any previous treatment with a poly adenosine diphosphate-ribose polymerase (PARP) inhibitor, including olaparib.
5. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
6. Patients receiving the following classes of inhibitors of cytochrome P450 3A4 (CYP3A4)

   * Azole antifungals
   * Macrolide antibiotics
   * Protease inhibitors
7. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
8. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, or any psychiatric disorder that prohibits obtaining informed consent.
9. Patients with a history of interstitial lung disease, inflammatory lung conditions, or severe chronic obstructive pulmonary disease (COPD) (FEV1<1litre or < 30% predicted). Patients with pneumonia within the previous 3 months.
10. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
11. Patients with oesophageal stent in-situ
12. Patients with myelodysplastic syndrome/acute myeloid leukaemia
13. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
14. Patients with known active hepatic disease (i.e., Hepatitis B or C).
15. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
16. Patients with uncontrolled seizures.
17. Concurrent uncontrolled medical illness, or other previous or current malignant disease likely to interfere with protocol treatments / comparisons
18. Age < 18
19. Any pregnant, lactating women or potentially childbearing patients not using adequate contraception (see section 3.4 for details of required contraception).
20. Previous chemotherapy or radiotherapy for oesophageal cancer
21. Metastatic disease apart from local lymph node disease which can be reasonably encompassed within the radiotherapy volume (total length of tumour and lymph node disease should be <10cm)
22. ECOG performance status >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of olaparib in combination with radical radiotherapy in patients with oesophageal cancer | 3 months post treatment
  MTD will be determined by the number of patients experiencing dose limiting toxicities (DLTs) in each treatment cohort, using a 3+3 dose escalation schedule. A DLT is determined as grade 4 oesophagitis or dysphagia, or any other grade 3 toxicity. DLTs will be assessed weekly during treatment (day -3 to week 5), 10-14 days after completing treatment, weekly for a further 3 weeks and 3 months after completing treatment.

SECONDARY OUTCOMES:
Overall toxicity profile of treatment (NCRI Common Toxicity Criteria for Adverse Effects V3) | Assessed at all study visits, up to 3 years post treatment.
  Toxicity of treatment will be assessed via collection of adverse events, categorised by the NCRI Common Toxicity Criteria for Adverse Effects (CTCAE) V3. Adverse event data will be collected continuously from screening, with patients seen weekly during their treatment, 10-14 days after treatment completion, weekly for 3 further weeks, 3 monthly until 1 year then 6 monthly until 3 years.
Olaparib compliance | At completion of olaparib treatment (end of week 5)
Radiotherapy (RT) compliance | At completion of RT treatment (end of week 5)
Local and overall treatment failure rate | 3 months
  This is defined as residual disease pathologically on endoscopic assessment & biopsy or progressive disease on CT scan of thorax and abdomen.
Exploration of blood and tissue borne pharmacodynamic markers to establish the biological efficacy of the addition of Olaparib to radiotherapy. | Up to 3 months post treatment
  * Endoscopic biopsy sample taken for analysis at screening & 3 months post treatment
  * Translational research blood samples taken at screening, weekly during treatment, at end of treatment visit & 3 months after treatment
  * Skin biopsy samples taken from within & outside irradiated field at week 4

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Jackson, Dr, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - Southampton General Hospital, Southampton